CLINICAL TRIAL: NCT05092646
Title: A Double-blind, Multi-Center, Prospective, Randomized Placebo-controlled Pilot Study Evaluating Intra-articular Injection of Axolotl Ambient Compared to Saline in Subjects With Ankle Osteoarthritis
Brief Title: Evaluating Intra-articular Injection of Axolotl Ambient Compared to Saline in Subjects With Ankle Osteoarthritis
Acronym: Phoenix
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Study stopped due to lack of enrollment
Sponsor: Axolotl Biologix (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CA-2021-01
Record Dates: First submitted 2021-10-08; First posted 2021-10-25 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Ankle Osteoarthritis
Keywords: Osteoarthritis, Biologic, Amniotic Fluid
MeSH Terms: conditions — Osteoarthritis | interventions — Saline Solution

STUDY DESIGN:
Intervention Model Description: Randomized, Placebo-controlled, Double-blinded
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Subjects, investigators, and outcome assessors will be blinded to the treatment allocation until completion of the 6-month follow-up visit.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Control Group (Placebo Comparator): Single dose, 2.0 mL of 0.9% normal saline, administered via intra-articular injection administered to the affected tibiotalar joint.
  Interventions: Drug: "Drug/Placebo: 0.9% Normal Saline"
- Investigational Group (Experimental): Biological/Vaccine: Axolotl Ambient
  Axolotl Ambient is an allogeneic amniotic intraarticular injection therapy consisting of a growth factor and cytokine-rich fluid derived from human amnion cells.
  Other Names:
  • CA20
  Interventions: Biological: Axolotl Ambient

INTERVENTIONS:
Biological: Axolotl Ambient — Axolotl Ambient is an allogeneic amniotic intra-articular injection therapy consisting of a growth factor and cytokine-rich fluid derived from human amnion cells.
  Other Names: CA20
  Arms: Investigational Group
Drug: "Drug/Placebo: 0.9% Normal Saline" — "Drug/Placebo: 0.9% Normal Saline"
  Arms: Control Group

SUMMARY:
A Double-blind, Multi-Center, Prospective, Randomized Placebo-controlled Pilot Study Evaluating Intra-articular Injection of Axolotl Ambient Compared to Saline in Subjects with Ankle Osteoarthritis. The goal of this pilot study and subsequent pivotal trial is to evaluate the safety and effectiveness of Axolotl Ambient intra-articular injection for ameliorating the pain and dysfunction associated with ankle OA.

DETAILED DESCRIPTION:
This pilot study is a double-blind multi-center, prospective, randomized, placebo-controlled trial. Upon randomization, patients will receive 1 intraarticular injection of the investigational product or control fluid. Follow-up will be conducted at 4 weeks, 3 and 6 months, with 6 months serving as the primary endpoint. The primary outcomes will consist of patient reported outcomes of pain and functional assessment by the physician, specific to the foot and ankle. Subjects will be monitored for an additional 6 months to establish safety over a 1-year follow-up and evaluate the durability of benefit.

ELIGIBILITY:
Inclusion Criteria:

1. Signed written informed consent
2. Willing to be randomized to either the investigational or control group
3. Male or female at least 18 years of age and less than 80
4. Clinical diagnosis of symptomatic tibiotalar (ankle) OA (primary idiopathic OA or post-traumatic OA), modified K-L grade 1-3a
5. One ankle is the most symptomatic lower extremity joint and the only lower extremity joint currently planned for treatment
6. Willing and able to comply with all study requirements including all postoperative clinical and radiographic evaluations
7. For women of childbearing potential (not post-menopausal for 12 months or surgically sterile), a urine pregnancy test with a negative result must be obtained at screening and on the day of procedure, prior to injection
8. Male and female trial participants must commit to adequate birth control (e.g., surgically sterilized, oral contraceptive, two methods of barrier birth control, or abstinence) through the final follow-up
9. Chronic ankle pain for ≥ 6 months
10. SAOS Pain score ≥ 30 and ≤ 80 and AOS Function score ≥ 30 and ≤ 80
11. Willing to discontinue all prescription and over-the-counter pain medications being used for ankle OA symptoms for the duration of the study, except for acetaminophen, which is not allowed for the 3 days preceding each scheduled follow-up visit and the day of the follow-up visit.

Exclusion Criteria:

1. Previously received intra-articular injections in the index joint of Axolotl Ambient, bone marrow aspirate concentrate (BMAC), platelet-rich plasma (PRP), or other biologic-based products within the last 12 months.
2. Modified K-L Grade 3b or 4 osteoarthritis of the index joint
3. Diagnosis of ipsilateral peri-articular arthritis (e.g. subtalar joint) that the investigator determines may significantly confound the study results
4. Received intra-articular hyaluronic acid injection in the index joint within the last 6 months
5. Received intra-articular steroid injection in the index joint within the last 3 months
6. Prior major surgical repair or reconstruction of the ankle that the investigator determines may significantly confound the study results
7. Baseline pain catastrophizing score ≥ 23
8. Any surgery of the index ankle within the last 12 months
9. Planned arthroscopy or other procedure on the ankle during the study
10. Bilateral ankle OA requiring treatment of both ankles
11. Pregnancy, breastfeeding, or woman of child-bearing potential not using adequate contraception
12. Bone deficit
13. Charcot foot disease
14. Radiographic evidence of open epiphyses
15. Systemic inflammatory condition
16. Substantial vascular insufficiency
17. Current treatment with anticoagulants
18. Deformity in coronal, axial or sagittal plane greater the 30°
19. Patients weighing less than 47 kg.
20. BMI greater than 45 kg/m2
21. Documented medical history of, or radiographic evidence of, a bone disease (e.g. severe osteoporosis or avascular necrosis) or other condition (e.g., osteolysis)
22. Comorbidity that would limit the ability to administer any functional measurements
23. Has at the time of injection, a systemic or local infection at the site of injection
24. Medical condition, serious intercurrent illness, or extenuating circumstance that, in the opinion of the Investigator, would preclude participation in the study or potentially decrease survival or interfere with ambulation or rehabilitation (e.g., history of transient ischemic attack, stroke or liver disease)
25. Known hypersensitivity to penicillin
26. Known allergy to phenol red
27. Currently receiving treatment with a drug known to interfere with bone or cartilage metabolism [e.g., systemic steroid therapy (topical steroid therapy is permissible), methotrexate]
28. Medical condition requiring radiation, chemotherapy or immunosuppression
29. Have an active history of malignancy (except for basal cell carcinoma of the skin)
30. Has a history of autoimmune disease known to affect bone or cartilage. Examples include spondyloarthropathies (e.g., ankylosing spondylitis, Crohn's disease, and ulcerative colitis), Juvenile Arthritis, rheumatoid arthritis, Grave's disease, and Hashimoto's thyroiditis
31. Has obvious or documented alcohol or illicit drug addictions
32. Is a prisoner in a correctional institution/facility
33. Actively involved in litigation or workman's compensation
34. Has participated in clinical studies evaluating investigational devices, pharmaceuticals or biologics within 6 months of randomization
35. Bedridden, confined to a wheelchair, or unable to walk 50 m without the help of a walker, crutches, or cane
36. Is currently taking prescription pain medication for any conditions other than ankle osteoarthritis.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-11-10 (Actual); Study Completion 2023-11-10 (Actual)

PRIMARY OUTCOMES:
Proportion of patients achieving Composite Clinical Success | 4 Weeks
  Changes from baseline to each follow-up timepoint (4 weeks, 3 and 6 months) will be calculated for each outcome metric and statistical significance of changes will be assessed through repeated measures ANOVA or a mixed effects model to accommodate missing data points. Two options (based on either AOS or FAOS scores) for CCS will be defined as:
  * Improvement in AOS (Pain and Function, independently) or FAOS (Pain and ADL, independently) subdomain scores of at least 20% from baseline
  AND
  * No medical or surgical intervention beyond allowed rescue medication
  AND
  * Absence of treatment-related SAEs
Proportion of patients achieving Composite Clinical Success | 3 Months
  Changes from baseline to each follow-up timepoint (4 weeks, 3 and 6 months) will be calculated for each outcome metric and statistical significance of changes will be assessed through repeated measures ANOVA or a mixed effects model to accommodate missing data points. Two options (based on either AOS or FAOS scores) for CCS will be defined as:
  * Improvement in AOS (Pain and Function, independently) or FAOS (Pain and ADL, independently) subdomain scores of at least 20% from baseline
  AND
  * No medical or surgical intervention beyond allowed rescue medication
  AND
  * Absence of treatment-related SAEs
Proportion of patients achieving Composite Clinical Success | 6 Months
  Changes from baseline to each follow-up timepoint (4 weeks, 3 and 6 months) will be calculated for each outcome metric and statistical significance of changes will be assessed through repeated measures ANOVA or a mixed effects model to accommodate missing data points. Two options (based on either AOS or FAOS scores) for CCS will be defined as:
  * Improvement in AOS (Pain and Function, independently) or FAOS (Pain and ADL, independently) subdomain scores of at least 20% from baseline
  AND
  * No medical or surgical intervention beyond allowed rescue medication
  AND
  * Absence of treatment-related SAEs

SECONDARY OUTCOMES:
Incidence of Adverse Events | Baseline (Day 0) to 12 Months
  An Adverse Event (AE) is any untoward medical occurrence, unintended disease or injury, or untoward clinical signs (including abnormal laboratory findings) in study subjects whether or not considered related to the investigational product. This definition includes events related to the investigational product or the comparator and events related to the procedures involved.
Symptoms, Quality of Life and Sports and Recreation subscales of the FAOS | Baseline (Day 0), 4 Weeks, 3 Months, 6 Months, and 12 Months
  The FAOS score was developed to reflect a foot and ankle version of the Knee Osteoarthritis Outcomes Score (KOOS). The FAOS score includes symptoms, quality of life and sports and recreation subscales.
Visual Analog Scale for average ankle pain and worst ankle pain | Baseline (Day 0), 4 Weeks, 3 Months, 6 Months, and 12 Months
  The Visual Analog Scale (VAS) is a measure of pain intensity. It is a continuous scale comprised of a horizontal visual analog scale anchored by two verbal descriptors (one for each symptom extreme).
EuroQOL-5 dimension-5 level quality of life scale | Baseline (Day 0), 4 Weeks, 3 Months, 6 Months, and 12 Months
  EQ-5D-5L is a self-completed health status questionnaire that assesses quality of life.
Pain Catastrophizing Scale | Baseline (Day 0), 4 Weeks, 3 Months, 6 Months, and 12 Months
  The pain catastrophizing scale (PCS) is a 13-item questionnaire that asks participants to grade each item on a 5-point scale.
Current Working Status | Baseline (Day 0), 4 Weeks, 3 Months, 6 Months, and 12 Months
  Percent of subject responses, for each of the following work status categories, by the treatment and control groups, at each timepoint.
  Current Working status, at each timepoint will be collected as:
  Not working, unrelated to ankle
  Not working, related to ankle
  Working with major limitations related to ankle
  Working without limitations related to ankle
Modified Kellgren and Lawrence Grade | Baseline (Day 0), 6 Months
  The modified Kellgren and Lawrence Grade (K-L Grade) classifies osteoarthritis using five grades based on evaluation of x-ray of the affected joint.

CONTACTS AND LOCATIONS:
Overall Officials: Robert S. Kellar, PhD, Study Director — Chief Science Officer (CSO); Aaron J. Tabor, PhD, CTBS, Study Director — V.P. of Clinical Operations
Locations (3):
- United States (3):
  - Injury Care Research, Boise, Idaho
  - Orthopedic Specialists of Louisiana, Shreveport, Louisiana
  - OrthoCarolina Foot and Ankle Institute, Charlotte, North Carolina

IPD SHARING:
Plan to Share IPD: No